CLINICAL TRIAL: NCT04367038
Title: The Impact of Different Acupressure Procedures Performed on the Hand During Labor on Endorphin Levels and Labor Pain Perception: A Randomised Controlled Trial
Brief Title: Endorphin at Labor Pain and Acupressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Serap ÖZTÜRK ALTINAYAK (Other)
Responsible Party: Sponsor-Investigator, Serap ÖZTÜRK ALTINAYAK, PhD, Academician, Tokat Gaziosmanpasa University
Organization: Tokat Gaziosmanpasa University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 25.09.2018-04/2
Record Dates: First submitted 2020-04-23; First posted 2020-04-29 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Labor Pain
Keywords: acupressure; labor pain; Midwifery; pregnant women; endorphins; warm acupressure; cold acupressure
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Warm Acupressure Procedure Group (Experimental): Latent phase Visual Analog Scale and Verbal Category Scale I given as pretest First venous blood sample taken Active phase The first warm acupressure procedure was performed for ten minutes on the Large Intestinal 4 energy meridian zone acupressure point on the non-dominant hand. This process was repeated three more times at one-hour intervals.
  Visual Analog Scale II and Verbal Category Scale II were measured at the end of the active phase Transition phase The second warm acupressure procedure was performed three times at one-hour intervals A 30-minute break was given Visual Analog Scale III and Verbal Category Scale III were performed Second venous blood sample taken
  Interventions: Other: Warm Acupressure, Cold Acupressure , Conventional Acupressure
- Cold Acupressure Procedure Group (Experimental): Latent phase Visual Analog Scale I and Verbal Category Scale I given as pretest First venous blood sample taken Active phase The first cold acupressure procedure was performed for ten minutes on the Large Intestinal 4 energy meridian zone acupressure point on the non-dominant hand. This process was repeated three more times at one-hour intervals.
  Visual Analog Scale II and Verbal Category Scale II were measured at the end of the active phase Transition phase The second cold acupressure procedure was performed three times at one-hour intervals A 30-minute break was given Visual Analog Scale III and Verbal Category Scale III were performed Second venous blood sample taken
  Interventions: Other: Warm Acupressure, Cold Acupressure , Conventional Acupressure
- Conventional Acupressure Group (Experimental): Latent phase Visual Analog Scale I and Verbal Category Scale I given as pretest First venous blood sample taken Active phase Conventional acupressure was performed for 30 minutes on the Large Intestinal 4 energy meridian zone acupressure point on the non-dominant hand. This process was repeated twice more at one-hour intervals.
  Visual Analog Scale II and Verbal Category Scale II were measured at the end of the active phase Transition phase The second conventional acupressure procedure was performed twice at one-hour intervals A 30-minute break was given Visual Analog Scale III and Verbal Category Scale III were performed Second venous blood sample taken
  Interventions: Other: Warm Acupressure, Cold Acupressure , Conventional Acupressure
- Control Group (No Intervention): Latent phase Visual Analog Scale I and Verbal Category Scale I given as pretest First venous sample taken Active phase
  No procedure other than the routine clinical practices were carried out. Visual Analog Scale II and Verbal Category Scale II were measured at the end of the active phase Transition phase No procedure other than the normal clinical routines was conducted Visual Analog Scale III and Verbal Category Scale III were performed. Second venous blood sample taken

INTERVENTIONS:
Other: Warm Acupressure, Cold Acupressure , Conventional Acupressure — Acupressure is non-invasive, safe and effective.
  Arms: Cold Acupressure Procedure Group; Conventional Acupressure Group; Warm Acupressure Procedure Group

SUMMARY:
This study was performed to determine the impact of different acupressure procedures, performed on women's hands during labor, on endorphin levels and labor pain perception.

The sample consisted of 140 pregnant women. The study was conducted with three experimental groups and one control group, each including 35 pregnant women. Conventional acupressure and warm and cold acupressure procedures were performed on the Large Intestinal 4 energy meridian zone acupressure point of the experimental group. No procedures were performed on the women in the control group. Data were collected using a "Personal Information Form", "Labor Intervention Follow-up Form", "Visual Analog Scale" and "Verbal Category Scale".

The comparison between the experimental and control groups indicated that the conventional acupressure procedure was effective in reducing labor pain and that the warm acupressure procedure increased endorphin levels.

ELIGIBILITY:
Inclusion Criteria:

* Being a primipara
* Having intact membranes
* No skin diseases (such as urticaria...),
* No use of narcotic drugs
* Having a term pregnancy
* Having a single fetus at vertex position
* Planning to have vaginal delivery
* Having contractions and ongoing regular augmentation
* Having recent augmentation starting periods
* Being in the latent phase (0-3 cm dilatation)
* Having no history of high-risk pregnancy
* Not using analgesic drugs to reduce pain during delivery
* Having no systemic and neurologic diseases
* Having no contraction anomaly (hypotonic or hypertonic contractions)

Exclusion Criteria:

Having any of the above criteria.

-

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2020-01-08 (Actual)

PRIMARY OUTCOMES:
labor pain | through study completion, an average of 1month
  pain scale
endorphin levels | through study completion, an average of 1month
  physiological parameter

CONTACTS AND LOCATIONS:
Overall Officials: Hava Özkan, PhD, Study Director — Atatürk University Faculty of Health Science, Department of Midwifery,
Locations (1):
- Health Research and Training Hospital of Tokat Gaziosmanpaşa University, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I want it published in a journal first.